CLINICAL TRIAL: NCT06917014
Title: A Randomized Controlled Study of Hysteroscopic "360°" Surgery for Improvement of Symptoms in Cesarean Scar Defects
Brief Title: Hysteroscopic "360°" Surgery for Improvement of Symptoms in Cesarean Scar Defects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Xiaowu Huang, Director of department, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-11-2331
Record Dates: First submitted 2025-03-25; First posted 2025-04-08 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cesarean Scar Defect
Keywords: Hysteroscopic "360°" Surgery; Cesarean Scar Defects

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 360° (Experimental): The interference of the experimental group is to resect the fibrotic inflamed tissue of the proximal and distal part of the niche, a high-frequency angled ball electrode was used to obtain focused coagulation of all residual inflamed tissue still present on the niche surface and on the cervical canal walls, focused electrocauterization with a ball electrode controlling any bleeding of the endocervical vessels.
  Interventions: Procedure: 360°
- traditional (Other): The interference of the control group is to resect the fibrotic tissue of the proximal of the niche, use angled ball electrode coagulation.
  Interventions: Procedure: traditional

INTERVENTIONS:
Procedure: 360° — reset the proximal and distal part of the niche, widely 360° coagulation to restore and change the shape and size of niche, and ultimately improve symptoms of patients.
  Arms: 360°
Procedure: traditional — reset the proximal part of the niche, and coagulation to restore and change the shape and size of niche, and ultimately improve symptoms of patients.
  Arms: traditional

SUMMARY:
Patients with symptomatic Cesarean Scar Defect (CSD) who are expected to undergo hysteroscopic surgery will be randomly divided into the traditional hysteroscopic "channelization" treatment group and the hysteroscopic "360 °" Surgery group of cesarean diverticulum, and the improvement of postoperative clinical symptoms of the two groups will be compared. To evaluate the effectiveness of the two surgical methods.

The purpose of this study was to evaluate the improvement of symptoms of women with symptomatic cesarean diverticulum through a high-quality randomized controlled study, in order to provide high-level evidence-based medical evidence for clinical treatment.

DETAILED DESCRIPTION:
1. Study Design：This is a prospective, randomized controlled trial.
2. Study population 120 patients diagnosed with Cesarean Scar Defect (CSD) will be prospectively recruited. Before the surgery all patients will undergo preoperative evaluations, including a detailed history of the menstrual pattern,any previous History of cesarean section, and reproductive history, as well as trans-vaginal ultrasonography and Three-dimensional SIS Ultrasound.
3. Randomization:

   Randomization was performed electronically using SPSS statistical software version 26.0 (SPSS, Inc., Chicago, IL,USA) by the investigator.120 recruited patients will be randomized to one of the two treatment groups by computer-generated numbers: the control group("channelization" group) and the experimental group("360°" group).
4. Surgical technique:

   Hysteroscopic surgery will be performed in a standardized manner.The procedure will be performed under general anesthesia. Ultrasonographic guidance will be routinely used.

   The interference of "360°" group (the experimental group) including 60 CSD patients ,With the vaginoscopic approach, the isthmocele was localized; a high-frequency 90°angled circular loop electrode and pure cutting current of 100 W were used to resect the fibrotic tissue of the proximal (step 1) and distal (step 2) part of the niche. The investigators performed resection not only of the fibrotic tissue underneath the niche but also of the inflamed tissue placed around the niche and on the opposite site (the so-called channel-like 360° endocervical ablation). A high-frequency angled ball electrode was used to obtain focused coagulation of all residual inflamed tissue still present on the niche surface and on the cervical canal walls (step 3); the aim of this step is to facilitate the re-epithelialization of the cervical canal walls by the paraphysiological endocervical epithelium. The procedure was ended by controlling any bleeding of the endocervical vessels by reducing the inflow and pressure of the distending medium and by focused electrocauterization with a ball electrode (step 4).while the interference of "channelization" group (the control group) , With the vaginoscopic approach, the isthmocele was localized; a high-frequency 90°angled circular loop electrode and pure cutting current of 100 W were used to resect the fibrotic tissue of the proximal perform intrauterine adhesiolysis with bipolar electric needle electrode, part of the scar tissue removed by electronic loop when it is necessary.A angled ball electrode was used to obtain focused coagulation of proliferating blood vessels, inflammatory tissue, and ectopic endometrium in the diverticulum.In both arms, the endometrium tissue was removed and sent to pathology, followed by immunohistochemical CD138 examination
5. Postoperative treatments All subjects will be treated with oral antibiotics for 3 days. Three-dimensional SIS Ultrasound will be carried out 3 months after the surgery.
6. Follow up:

   Follow-up styles: the doctor's outpatient review, patients fill in questionnaires,telephone, WeChat and so on.

   Follow-up time:3 months and 6 months after the operation. Follow-up contents: the data measured by 3D-SIS,At the same time, the endometrium was taken again for immunohistochemical CD138 examination. Assessed the improvement of symptoms, including the improvement of prolonged menstrual period, the improvement of heavy menstruation, and the patient's postoperative satisfaction.
7. Consent： All subjects will be given a detailed explanation of the study and sufficient time to consider their participation. A written consent form will be signed by the patient and retained in the records.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgical adaptation: changes in menstruation after cesarean section (prolonged menstrual period)
* No surgical contraindications;
* Age 18-45 years old;
* The thickness of residual muscle layer measured by ultrasound is greater than or equal to 2.5mm;
* Patients with symptoms that have not improved significantly for more than 1 month after oral short-acting contraceptive cycle treatment or who strongly require surgery;
* Understand and agree to the research plan.

Exclusion Criteria:

* Patients with other diseases that may cause abnormal uterine bleeding (including endometrial polyps, endometrial hyperplasia, submucosal myoma, etc.) indicated by two-dimensional ultrasound
* There are contraindications of surgery: such as severe internal and surgical complications, pregnancy, reproductive tract infection, malignant tumor;

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-05-16 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Symptom change rate | 6 months after surgery
  Rate of change in abnormal bleeding before and after the operation

SECONDARY OUTCOMES:
Ultrasound measurement values | 3 months after surgery
  Ultrasound measurement values before and after the operation，include residual muscle thickness;length of cesarean scar defects;width of cesarean scar defects;height of cesarean scar defects

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casadio P, Gubbini G, Morra C, Franchini M, Paradisi R, Seracchioli R. Channel-like 360 degrees Isthmocele Treatment with a 16F Mini-Resectoscope: A Step-by-step Technique. J Minim Invasive Gynecol. 2019 Nov-Dec;26(7):1229-1230. doi: 10.1016/j.jmig.2019.04.024. Epub 2019 May 3. PMID 31059782
- [Background] Casadio P, Raffone A, Alletto A, Filipponi F, Raimondo D, Arena A, La Rosa M, Virgilio A, Franceschini C, Gubbini G, Franchini M, Paradisi R, Lenzi J, Travaglino A, Mollo A, Carugno J, Seracchioli R. Postoperative morphologic changes of the isthmocele and clinical impact in patients treated by channel-like (360 degrees ) hysteroscopic technique. Int J Gynaecol Obstet. 2023 Jan;160(1):326-333. doi: 10.1002/ijgo.14387. Epub 2022 Aug 23. PMID 35929843
- [Background] Zhang NN, Wang GW, Yang Q. Endoscopic Treatment of Previous Cesarean Scar Defect in Women with Postmenstrual Bleeding: A Retrospective Cohort Study. J Invest Surg. 2021 Oct;34(10):1147-1155. doi: 10.1080/08941939.2020.1766161. Epub 2020 May 13. PMID 32404009
- [Background] Shapira M, Mashiach R, Meller N, Watad H, Baron A, Bouaziz J, Cohen SB. Clinical Success Rate of Extensive Hysteroscopic Cesarean Scar Defect Excision and Correlation to Histologic Findings. J Minim Invasive Gynecol. 2020 Jan;27(1):129-134. doi: 10.1016/j.jmig.2019.03.001. Epub 2019 Mar 8. PMID 30858053
- [Background] He Y, Zhong J, Zhou W, Zeng S, Li H, Yang H, Shan N. Four Surgical Strategies for the Treatment of Cesarean Scar Defect: A Systematic Review and Network Meta-analysis. J Minim Invasive Gynecol. 2020 Mar-Apr;27(3):593-602. doi: 10.1016/j.jmig.2019.03.027. Epub 2019 Nov 5. PMID 31698049